CLINICAL TRIAL: NCT03321409
Title: The Validation of the Somatic Symptom Scale China (SSS-CN) for Assessing Somatic Symptom Burden and Its Utility in Patients With Suspected Coronary Artery Disease
Brief Title: Assessment of Somatic Symptom Burden
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Peking University People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Other Study IDs: SSS201709
Record Dates: First submitted 2017-10-03; First posted 2017-10-25 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Somatization Disorder
Keywords: Somatic symptom; SSS-CN; PHQ-15; Suspected CAD; Coronary angiography
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The general population: People who take the physical examination in Renji Hospital between 18 to 80 years old without any previously confirmed serious medical conditions or mental disorders.
  Interventions: Diagnostic Test: The general population
- The patients with suspected CAD: Patients with suspected CAD between 18 to 80 years old without any previously confirmed serious medical conditions or mental disorders.
  Interventions: Diagnostic Test: Patients with suspected CAD

INTERVENTIONS:
Diagnostic Test: The general population — After recruiting participants, collecting the baseline data, the SSS-CN and PHQ-15 will be carried out. Then validating the reliability, validity of the SSS-CN will be compared with the PHQ-15.
  Other Names: SSS-CN and PHQ-15 questionnaire
  Groups: The general population
Diagnostic Test: Patients with suspected CAD — In patients with suspected CAD, after recruiting participants, collecting the baseline data, the SSS-CN and PHQ-15 will be carried out before undergo coronary angiography. Then the prevalence of somatic symptoms will be investigated.
  Other Names: SSS-CN and PHQ-15 questionnaire before coronary angiography
  Groups: The patients with suspected CAD

SUMMARY:
The Patient Health Questionnaire-15 (PHQ-15) is a frequently used questionnaire to assess somatic symptom burden. The Somatic Symptom Scale China (SSS-CN) was recently developed as a comprehensive self-report instrument in assessing somatic symptom burden, but its assessment value has not yet been widely tested in a nationwide. The study aims to investigate the reliability of the SSS-CN, to validate discriminate validity and factorial validity, and to investigate its utility in patients with suspected coronary artery disease (CAD) based on multi-centers inpatients.

DETAILED DESCRIPTION:
Somatic symptoms are prevalent in kinds of medical conditions and mental disorders. Since they are associated with decreased quality of life, increased psychological distress, and increased use of health care services, the assessment of somatic symptom burden is essential in evidence based patient care and research. The Patient Health Questionnaire-15 (PHQ-15) is a frequently used questionnaire to assess somatic symptom burden, but in which there are not any mental symptoms listed. Recently, we developed the Somatic Symptom Scale China (SSS-CN) which includes common mental symptoms and more comprehensive somatic symptoms to assess somatic symptom burden, but its assessment value has not yet been widely tested.

The aim of our study is to investigate the reliability and validity of the SSS-CN compared with the PHQ-15. We also try to use the SSS-CN to investigate the prevalence of somatic symptoms in patients with suspected coronary artery disease (CAD) based on multi-centers inpatients.

ELIGIBILITY:
Inclusion Criteria:

1. People who take the physical examination in Renji Hospital.
2. Patients with suspected CAD.

Exclusion Criteria:

1. People who have been previously confirmed serious medical conditions.
2. People who have been previously confirmed serious mental disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects are enrolled into 2 cohorts between September 2017 and June 2019. The cohorts are divided as the general population and the patients with suspected CAD.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The score of the SSS-CN in the general population | Within 24 hours after collecting the scale.
  To investigate the cutoff, reliability and validity of the SSS-CN according to the score.
  The Somatic Symptom Scale China (SSS-CN) is developed to assess somatic symptom burden, which includes 20 items. Each item represents an organ discomfort and is rated as 1 ("not at all"), 2 （"mild"）, 3（"moderate"）， or 4 ("severe"). In determining the SSS-CN score, the total score is summarized from the 20 items, rendering ranges from 20 to 80 (higher scores represent the more severe somatic symptom burden).

SECONDARY OUTCOMES:
Number of participants with somatic burden in suspected CAD patients | Within 24 hours after the coronary angiography.
  To validate the utility of SSS-CN and investigate the prevalence of somatic burden in patients with suspected CAD as assessed by SSS-CN.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China